CLINICAL TRIAL: NCT07295483
Title: To Analyze the Determining Factors in the Evolution of Subjects Diagnosed With Long COVID at Four Years of Follow-up. BioICOPER Follow-up Study.
Brief Title: Predictors of Long-Term Evolution in Long COVID; 4-Year Follow-Up. (BioICOPER Follow-up Study)
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto de Investigación Biomédica de Salamanca (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: BioICOPER Follow-up Study
Record Dates: First submitted 2025-11-20; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Persistent COVID Condition
Keywords: Post-acute COVID syndrome; Vascular aging; Proteomics; Biomarkers; Machine learning; Persistent COVID; Artificial Intelligence
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — Serum and plasma samples for proteomic and biomarker analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BioICOPER Long COVID Cohort: Adults previously enrolled in the BioICOPER study with a clinical diagnosis of long COVID.
  Interventions: Other: BioICOPER Long COVID Cohort

INTERVENTIONS:
Other: BioICOPER Long COVID Cohort — This observational cohort includes 400 adult participants previously enrolled in the baseline BioICOPER study (2021-2023), who had a confirmed diagnosis of long COVID (persistent COVID-19) according to WHO criteria.
  Participants will undergo a comprehensive four-year follow-up assessment to evaluate clinical evolution, vascular function, and biological markers of disease persistence and recovery.
  There is no intervention assigned by the investigators - participants will continue their usual medical care.
  The study will observe natural disease progression and its association with biomarkers, vascular measurements, and lifestyle factors.

SUMMARY:
Long COVID (persistent COVID) represents a major global health challenge due to its high prevalence (approximately 7%), significant impact on quality of life, and socioeconomic burden. Despite extensive research, diagnostic tools to objectively identify or predict long COVID evolution are still lacking.

The BioICOPER Follow-up Study aims to analyze the influence of biomarker evolution on clinical symptomatology (particularly chronic fatigue) and vascular health after four years of follow-up among 400 participants previously included in the original BioICOPER cohort.

Advanced proteomic analysis, vascular function assessment, and machine-learning-based predictive modeling will be used to identify biomarkers associated with disease progression, stratified by sex. This project will contribute to personalized clinical management of long COVID and improved diagnostic and therapeutic strategies in primary care.

DETAILED DESCRIPTION:
The study includes a citizen participation component through the IBSAL Citizen Committee for review and dissemination of results. A prospective observational cohort study following 400 adults with a confirmed diagnosis of long COVID, previously enrolled in the BioICOPER baseline study.

Participants will undergo reevaluation four years after their initial inclusion, assessing:

* Clinical symptoms (fatigue, dyspnea, sleep, cognition, nutrition, frailty).
* Lifestyle factors (physical activity, diet, alcohol and tobacco use).
* Vascular structure and function using carotid ultrasound, pulse wave velocity (SphygmoCor®, Vasera®), and retinal imaging.
* Proteomic profiling and quantification of SARS-CoV-2 N and S proteins using ELISA and mass spectrometry.
* Predictive modeling using artificial intelligence (AI) and bioinformatics methods (ESALAB group).

The study will identify biological, vascular, and behavioral determinants of long COVID progression, aiming to build predictive models to support personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old.
* Confirmed previous SARS-CoV-2 infection.
* Diagnosis of long COVID according to WHO criteria.
* Participation in the baseline BioICOPER study.
* Signed informed consent for re-evaluation.

Exclusion Criteria:

* Acute illness preventing participation.
* Cognitive or physical impairment limiting data collection.
* Withdrawal of informed consent.
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults previously enrolled in the BioICOPER study with a clinical diagnosis of long COVID.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression of vascular stiffness measured by carotid-femoral pulse wave velocity (cfPWV) | From baseline to 48-month follow-up
  Carotid-femoral pulse wave velocity will be assessed as the gold-standard measure of arterial stiffness, using the SphygmoCor® system. The study will evaluate the longitudinal change in cfPWV between baseline (BioICOPER inclusion) and the 4-year follow-up visit, in order to determine whether long COVID is associated with accelerated vascular aging.

SECONDARY OUTCOMES:
Change in Fatigue Severity Score (FSS) | From baseline to 4-year follow-up.
  Fatigue assessed using a validated fatigue scale (Fatigue Severity Scale, FSS). The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue on you. The FSS is a short questionnaire that requires the patient to rate their level of fatigue. The FSS questionnaire contains nine statements that rate the severity of their fatigue symptoms. the patient needs to read each statement and circle a number from 1 to 7, based on how accurately it reflects their condition during the previous week and the extent to which they agree or disagree that the statement applies to them.
  A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement.
  The goal of this outcome is to determine how fatigue severity evolves and its association with biomarkers and vascular parameters.
Change in Health-Related Quality of Life (EQ-5D-5L or SF-36) | From baseline to 4 years.
  EQ-5D-5L is a health-related quality of life survey that uses five questions, each with five severity levels, to measure health status across the dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Health state profile: A person's answers create a five-number profile that describes their current health state.
  Scoring: This profile can be used to calculate a single index score that represents health-related quality of life. This score ranges from 0 (death) to 1 (full health).
  It assesses eight health concepts: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
  The SF-36 survey grades health by scoring responses on eight different health domains, which are then converted to a 0-100 scale where higher scores indicate better health. A score of 100 represents the best possible health in that category, while 0 represents the worst.
Change in Cognitive Function (Montreal Cognitive Assessment, MoCA) | Baseline to 4 years
  Evaluate cognitive impairment associated with long COVID using the Montreal Cognitive Assessment, which is a 10-minute screening test used to detect mild cognitive impairment in adults. It is a 30-point test that evaluates several cognitive domains, including memory, attention, language, visuospatial skills, executive functions, and orientation. A score of 26 or above is considered a normal result, while lower scores may indicate some level of cognitive dysfunction. The goal of this assesment is to identify determinants of neurocognitive persistence or recovery.
Change in Physical Activity (WHO Physical Activity Questionnaire + 7-day pedometer readings) | Baseline to 4 years.
  Objectively and subjectively measure physical activity levels using both WHO Physical Activity Questionnaire and 7-day pedometer readings. The WHO Physical Activity Questionnaire is a 16 question instrument that assesses physical activity participation in three domains (activity at work, travel to and from places, and recreational activities) as well as sedentary behavior. Physical activity may include planned activity such as walking, running, basketball, or other sports. Physical activity may also include other daily activities such as household chores, yard work, walking the dog, etc. The use of the pedometer only completes the questionnaire, hence both variables need to be meassured simultaneously and interpret them together in order to determine changes in physical activity.
Change in Adherence to the Mediterranean Diet (PREDIMED Questionnaire) | Baseline to 4 years.
  Evaluate diet quality and its relation to metabolic and vascular outcomes. The PREDIMED questionnaire is a screening tool used in the PREDIMED study to assess adherence to the Mediterranean diet. The most common version is a 14-point questionnaire that asks about frequency of consumption of certain foods like olive oil, nuts, fruits, vegetables, and fish, and the limited intake of red meat, butter, and sugary drinks. Participants receive a score of 0 or 1 for each question, and the total score is used to classify their diet as low, moderate, or high in Mediterranean adherence. The goal of this outome is to assess dietary influence on systemic inflammation, endothelial function, and metabolic health.
Change in Body Composition (InBody 230 Bioimpedance Analysis) | Baseline to 4 years.
  The InBody 230 Bioimpedance Analysis is a non-invasive test that measures body composition by sending a mild electrical current through the body. It uses a technique called segmental multifrequency bioelectrical impedance to provide detailed information on body fat, skeletal muscle mass, and body water in the torso, arms, and legs. This analysis offers a more comprehensive picture of your health than a standard scale, providing data like Basal Metabolic Rate (BMR) and Body Mass Index (BMI). The goal od this outcome is to explore links between body composition and cardiovascular risk in long COVID.
Change in Biomarkers of Endothelial and Inflammatory Activity | Baseline to 4 years
  This Outcome Measure reflects a single assessment in which multiple plasma biomarkers (e.g., ICAM-1, VCAM-1, Endothelin-1, TNF-α, IL-10, and additional cytokines) are quantified within the same measurement framework. All biomarkers are measured using ELISA and proteomic techniques and reported in consistent concentration units (e.g., pg/mL or ng/mL) as appropriate for each assay. Although multiple biomarkers are included, they represent components of one integrated biomarker panel evaluating endothelial and inflammatory activity. No aggregation of different units is performed; instead, each biomarker's concentration is reported separately under this single Outcome Measure to characterize molecular pathways involved in long-term vascular and inflammatory changes in long COVID.
Change in Proteomic Profiles | 4 years
  Analysis of proteomic profiling of serum/plasma using advanced mass spectrometry to identify proteins related to fatigue, inflammation, and vascular aging to discover predictive biomarkers for persistent symptoms and disease progression.
SARS-CoV-2 Protein Quantification (N and S Proteins) | 4 years
  In order to explore persistence of viral antigens and relationship with ongoing symptoms and vascular damage, plasma will be qualified using ELISA.
AI-Based Predictive Model Performance | Baseline to 4 years.
  To develop and validate AI-based tools for risk stratification and personalized management using supervised learning (Random Forest, XGBoost, Neural Networks) trained on 70% of the cohort, validated on 30%. The machine learning models will combine clinical, vascular, and proteomic variables to predict disease trajectory.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Angel Gomez Marcos, MD, PhD, Principal Investigator — Centro Asistencial Universitario de Salamanca (CAUSA)
Locations (1):
- Av. de Portugal 83. Planta 2, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
Anonymized datasets and analytic code will be available upon reasonable request, following approval by the Ethics Committee and IBSAL data governance board.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available starting 12 months after publication of primary results and for a minimum of 5 years thereafter.
Access Criteria: Sharing Access Criteria: Qualified researchers with a methodologically sound proposal, as determined by the study steering committee, will be able to access the data. Requests should be directed to the study PI. A data access agreement will be required.